CLINICAL TRIAL: NCT04591860
Title: A Prospective Randomised Multi - Center Trial on the Repair of Large Hiatal Hernias With Sutures Versus Pledgeted Sutures Versus Absorbable Mesh
Brief Title: A Prospective Randomised Multi - Center Trial on the Repair of Large Hiatal Hernias: Absorbable Mesh vs. Pledgeted Sutures vs. Sutures Only
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paracelsus Medical University (Other)
Collaborators: Medical University Innsbruck (Other); Medical University of Vienna (Other); Krankenhaus Barmherzige Schwestern Linz (Other); Elisabethinen Hospital (Other)
Responsible Party: Principal Investigator, Michael Weitzendorfer, MD, Dr. Michael Weitzendorfer, PhD, Paracelsus Medical University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Phasix™ST - Austria
Record Dates: First submitted 2020-09-17; First posted 2020-10-19 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Hiatal Hernia
Keywords: hiatal hernia; pledgets; mesh; hernia recurrence
MeSH Terms: conditions — Hernia, Hiatal | interventions — Laparoscopy

STUDY DESIGN:
Intervention Model Description: The primary objective of the present trial is to compare the hiatal hernia recurrence rate between three different methods of cruroplasty in large hiatal hernias: hiatal closure with sutures versus pledgeted sutures versus absorbable mesh (Phasix™ST mesh).
  The study includes patients who are scheduled to undergo laparoscopic or robot-assisted surgery for a large symptomatic hiatal hernia. A large hiatal hernia is defined as > 5cm in manometry or gastroscopy or at least 1/3 of the stomach lying intrathoracically. The primary study endpoint is defined as the hernia recurrence rate, objectively assessed by gastroscopy. After inclusion in the study, patients will be followed up 6 months, 1 year, 3 years and 5 years after the operation using standardized questionnaires and gastroscopy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sutures only (Active Comparator): Patients with a large hiatal hernia undergo the cruroplasty with sutures only.
  A large hiatal hernia is defined as > 5cm in manometry or gastroscopy or at least 1/3 of the stomach lying intrathoracically.
  Interventions: Device: Laparoscopic or robot-assisted hiatal closure (sutures only vs. absorbable mesh vs. pledgeted sutures) and fundoplication according to Toupet
- Absorbable Mesh (Active Comparator): Patients with a large hiatal hernia undergo the cruroplasty with mesh implantation.
  A large hiatal hernia is defined as > 5cm in manometry or gastroscopy or at least 1/3 of the stomach lying intrathoracically.
  Interventions: Device: Laparoscopic or robot-assisted hiatal closure (sutures only vs. absorbable mesh vs. pledgeted sutures) and fundoplication according to Toupet
- Pledgeted sutures (Active Comparator): Patients with a large hiatal hernia undergo the cruroplasty with pledgeted sutures.
  A large hiatal hernia is defined as > 5cm in manometry or gastroscopy or at least 1/3 of the stomach lying intrathoracically.
  Interventions: Device: Laparoscopic or robot-assisted hiatal closure (sutures only vs. absorbable mesh vs. pledgeted sutures) and fundoplication according to Toupet

INTERVENTIONS:
Device: Laparoscopic or robot-assisted hiatal closure (sutures only vs. absorbable mesh vs. pledgeted sutures) and fundoplication according to Toupet — Patients are scheduled to undergo laparoscopic or robot-assisted surgery for a large symptomatic hiatal hernia.The hiatal closure will be done with sutures, pledgeted sutures or absorbable mesh (Phasix™ST mesh). After cruroplasty a fundoplication according to Toupet will be done additionally.

SUMMARY:
A prospective randomised multi - center trial on the repair of large hiatal hernias with sutures versus pledgeted sutures versus absorbable mesh

The primary objective of the present trial is to compare the hiatal hernia recurrence rate between three different methods of cruroplasty in large hiatal hernias: hiatal closure with sutures versus pledgeted sutures versus absorbable mesh (Phasix™ST mesh).

The duration of the study is not limited and depends on the number of cases planned. After enrollment in the study, patients will be followed - up with standardized questionnaires and gastroscopy at 6 months, 1 year, 3 years and 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a large hiatal hernia - admitted for surgery (laparoscopic / robot-assisted)
* Written informed consent
* ≥ 18 years of age
* Hiatal hernia documented by barium x-ray and/or gastroscopy and/or manometry by one or more of the following criteria:

  * > 5cm hiatal hernia
  * 1/3 of the stomach in the thorax

Exclusion Criteria:

* Lack of patient consent for study participation
* Lack of consent to study due to linguistic or mental incomprehension
* Patients in poor general condition (lack of anesthesia ability)
* Pregnancy
* Prior surgery on the stomach or gastroesophageal junction
* Simultaneous surgery because of another illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Hiatal hernia recurrence rate | 6 months, 1 year, 3 years and 5 years after surgery
  Hiatal hernia recurrence rate documented by gastroscopy

SECONDARY OUTCOMES:
Quality of Life evaluated by questionnaire | Prior to surgery; 6 months, 1 year, 3 years and 5 years after surgery
  Quality of Life measured by Gastrointestinal Quality of Life Index (GIQLI)
Symptoms related to Gastroesophageal Reflux Disease (GERD) | Prior to surgery; 6 months, 1 year, 3 years and 5 years after surgery
  Typical and atypical GERD symptoms assessed by the Symptom Check List (SCL) in units of a scale.
Primary extraesophageal GERD symptoms related to Gastroesophageal Reflux Disease (GERD) | Prior to surgery; 6 months, 1 year, 3 years and 5 years after surgery
  Primary atypical GERD symptoms assessed by the Reflux Symptom Index (RSI - Score) in units of a scale
Postoperative complications | 6 months, 1 year, 3 years and 5 years after surgery
  Short - term and long - term complications after treatment
Length of hospital stay | up to 90 days
  Length of hospital stay and mortality rates
Predictive parameters for treatment response or failure I | Prior to surgery; 6 months, 1 year, 3 years and 5 years after surgery
  Weight (in kilograms)
Predictive parameters for treatment response or failure II | Prior to surgery; 6 months, 1 year, 3 years and 5 years after surgery
  Height (in meters)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koch O, von Rahden BHA, Wykypiel H, Schoppmann SF, Fugger R, Rosanelli G, Emmanuel K, Weitzendorfer M. [Planning and Design of a Prospective Randomised Multi-Centre Trial on the Repair of Large Hiatal Hernias with Sutures vs. Pledgeted Sutures vs. Absorbable Mesh]. Zentralbl Chir. 2021 Apr;146(2):204-209. doi: 10.1055/a-1369-9694. Epub 2021 Feb 10. German. PMID 33567462